CLINICAL TRIAL: NCT07070466
Title: A Single-Arm, Phase II Study of Ivonescimab in Combination With FOLFOX in Advanced HER2 Negative Gastroesophageal Adenocarcinomas
Brief Title: Ivonescimab in Comb. With FOLFOX in Advanced HER2 Neg. GEA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Principal Investigator, Samuel J. Klempner, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-327
Record Dates: First submitted 2025-06-14; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Stomach Cancer Stage IV; Esophagus Cancer; Stomach Cancer
Keywords: stomach cancer; esophageal cancer; Phase 2; Immunotherapy
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ivonescimab plus FOLFOX (Experimental): Ivonescimab will be given once every 2 weeks into your vein (by intravenous infusion) over about 60 minutes. For the first treatment ivonescimab will be given alone with no chemotherapy.
  FOLFOX is a combination of 5-fluorouracil, oxaliplatin, and leucovorin. Starting Cycle 2 on beyond FOLFOX will be given after ivonescimab once every 2 weeks into your vein (intravenously). Some may be given over a shorter period of time (as short as approximately 1 minute) and others up to approximately 120 minutes.
  Ivonescimab in combination with FOLFOX will be given for up to 2 years as long as no serious side effects and disease does not worsen.
  Interventions: Drug: Ivonescimab; Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Drug: Ivonescimab — Humanized immunoglobulin G1 monoclonal antibody
Drug: 5-Fluorouracil — Nucleoside metabolic inhibitor
Drug: Oxaliplatin — Platinum-based drug and organoplatinum complex
Drug: Leucovorin — 5-formyl derivative of tetrahydrofolic acid

SUMMARY:
This is a single arm, open-label, phase II trial investigating the combination of ivonescimab with standard FOLFOX chemotherapy in 1L therapy for HER2- GEA.

DETAILED DESCRIPTION:
This is a single arm, open-label, non-randomized multi-institution phase II trial of the anti-PD-1 x VEGR bispecific antibody ivonoescimab in combination with standard 5-fluorouracil (5FU) and oxaliplatin as first line therapy in patients with locally advanced unresectable or metastatic HER2 negative (HER2-) gastroesophageal adenocarcinomas. The primary hypothesis is that the combination of dual VEGF and PD-1 targeting with standard 5FU/oxaliplatin (FOLFOX) will overcome intrinsic immunotherapy resistance and increase the objective response rate (ORR) and progression free survival (PFS) in frontline gastroesophageal adenocarcinomas (GEA). The goal is to determine the efficacy of this combination as measured by 6-month PFS rate and confirm the safety and tolerability in this target population.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologically confirmed diagnosis of adenocarcinoma of the esophagus, gastroesophageal junction, stomach. Squamous cell tumors are excluded. Patients with locally tested HER2 positive tumors (HER2+) tumors are excluded.
* Participants must have disease that can be evaluated radiographically. This includes disease that may be measurable or non-measurable as per RECIST version 1.1.
* Patients may not have received prior therapy for Stage IV disease. Patients may have received prior adjuvant therapy if more than 6 months have elapsed between the end of adjuvant therapy and registration.
* Age ≥18 years old. Because there is no dosing or adverse event data for ivonescimab with FOLFOX in participants <18 years of age, children are excluded from this study.
* ECOG Performance status of 0-2
* Participants must meet the following organ and marrow function as defined below:

  1. absolute neutrophil count ≥1,500/mcL
  2. hemoglobin > 9.0 g/dL
  3. platelets ≥100,000/mcL
  4. total bilirubin ≤ 1.5x institutional upper limit of normal (ULN). For patients with liver metastases or confirmed/suspected Gilbert syndrome, TBIL ≤3 × ULN
  5. AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN. For patients with liver metastases, AST and ALT ≤ 5 × ULN
  6. Creatinine ≤ institutional ULN OR glomerular filtration rate (GFR) ≥50 mL/min.
  7. Urine protein < 2+ or 24-hour protein quantification < 1.0 grams.
  8. Coagulation: prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 × ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (unless abnormalities are unrelated to coagulopathy) This applies only to patients who are not on therapeutic anti-coagulation. Patients receiving therapeutic anti-coagulation should be on a stable dose.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with brain metastases (active brain metastases) or leptomeningeal disease are not eligible. Patients with treated brain metastases who are off systemic steroids > 2 weeks and have documented radiographic stability over 4 weeks since initial brain metastasis diagnosis may be considered in discussion with the overall principal investigator.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The effects of ivonescimab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Contraception should continue for 9 months from the last dose of any study medication.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 9 months after completion of ivonescimab administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment with a PD-1 or PD-L1 inhibitor is exclusionary unless this therapy was completed > 6 months prior to the time of enrollment as part of adjuvant therapy.
* Major surgical procedures or serious trauma within 4 weeks prior to randomization, or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to randomization.
* Participants who have not recovered from adverse events due to prior adjuvant anti-cancer therapy except for alopecia or peripheral neuropathy grade 1 or less.
* Participants who are receiving any other investigational agents for this condition are not eligible.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ivonescimab. Patients with prior oxaliplatin and/or 5FU allergic reactions during adjuvant therapy are allowed if they have undergone prior desensitization with allergy and documented tolerance at standard dosing after desensitization.
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with ivonescimab. These potential risks may also apply to other agents used in this study.
* History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to randomization.
* Clinically significant hypertension with systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy.
* History of any grade arterial thromboembolic event, venous thromboembolic event of Grade 3 and above as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 12 months prior to randomization.
* Participants with a documented history of impaired wound healing are excluded.
* Participants with a history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Participants with uncontrolled intercurrent illness that would interfere with ability to participate in the opinion of the treating investigator.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 2) or unstable vascular disease (eg, aortic aneurysm at risk of rupture, Moyamoya disease) that required hospitalization within 12 months prior to randomization, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia).
* Subjects with any condition requiring systemic treatment with either corticosteroids (>2mg daily dexamethasone equivalent) or other immunosuppressive medications within 14 days of treatment. Premedication for hypersensitivity reactions (e.g. to contrast for CT or gadolinium for MRI) is allowed.
* Active systemic infection requiring intravenous antibiotics or intravenous monoclonal antibody treatments within 7 days of cycle 1 day 1.
* Participants with a known history of Human Immunodeficiency Virus (HIV) infection are excluded unless they meet all of the following criteria:

  * Stable antiretroviral therapy (ART) for at least 12 weeks prior to enrollment
  * No history of AIDS-defining conditions.
  * CD4+ T-cell count ≥ 350 cells/mm³ at screening
  * HIV viral load ≤ 50 copies/mL at screening.
  * No significant comorbidities associated with HIV infection that could interfere with the safety or efficacy of the investigational treatment.
  * No concurrent use of prohibited medications that may interfere with the study drug or cancer therapy
* History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to randomization, including but not limited to:

  * Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots). Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed.
  * Nasal bleeding /epistaxis (bloody nasal discharge is allowed)
  * Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to randomization is not allowed. The use of full-dose anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits according to the medical standard of the enrolling institution.
* History of non-infectious pneumonitis requiring therapy within 4 weeks of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
6-month progression free survival rate | From the start of treatment (Cycle 1, day 1) to first documented disease progression or date of death from any cause. Status at 6-months after starting treatment will be reported.
  The primary endpoint is to estimate the 6-month progression free survival rate for the combination of ivonescimab in combination with FOLFOX in frontline GEA adenocarcinomas. Progression is defined as measured from the start of the treatment with ivonescimab to the date of either documentation of disease progression or death. Progression of disease is defined per RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Incidence and Severity of Treatment-Emergent Adverse Events | From baseline until up to 90-days after end of study.
  Assessed using NCI Common Terminology for Adverse Event (CTCAE) version 5.0. All participants will be followed and assessed for safety and tolerability of the protocol therapy.
Objective Response Rate | From baseline until end of study or death, whichever comes first for up to 5 years.
  The percentage of participants that have a partial response or complete response.
Overall Clinical Benefit | From the baseline start of treatment to the date to first documented disease progression or date of death from any cause, whichever comes first for up to 5 years.
  This is defined by stable disease (SD), complete response rate (CR), or partial response (PR) assessed by RECISTv1.1. They will be summarized using binomial proportions along with exact 95% CI.
Median Progression Free Survival and Overall Survival | From baseline start of treatment to first documented disease progression or date of death from any cause, whichever comes first for up to 5 years.
  Median progression free survival is the length of time during treatment and after treatment to disease progression or death. Overall survival is the time from start if treatment to death due to any cause. The Kaplan-Meier method will be used to estimate median progression free survival and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klempner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber/Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to [sklempner@mgb.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation